CLINICAL TRIAL: NCT00893347
Title: Prevention of Persistent Post-concussion Syndrome With Cognitive-behavioural Therapy in At-risk Patients
Brief Title: An Intervention Program to Reduce to the Risk of Persistent Symptoms After Concussion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H08-02595
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2012-11

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild traumatic brain injury; Concussion; Post-Concussion Syndrome; Cognitive-Behavioural Therapy
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual
- II (Experimental): Treatment as usual + cognitive-behavioural therapy
  Interventions: Behavioral: Treatment as usual; Behavioral: Cognitive-behavioural therapy

INTERVENTIONS:
Behavioral: Treatment as usual — Single session with early intervention coordinator for assessment, education about mild traumatic brain injury, and recommendations for symptom management.
Behavioral: Cognitive-behavioural therapy — 6-session manualized cognitive-behavioural therapy protocol designed to prevent persistent post-concussion syndrome
  Arms: II

SUMMARY:
This study investigates how well a new therapy program prevents persistent symptoms (e.g., headaches, fatigue, irritability, etc.) after concussion. The program involves examining beliefs about concussion and learning healthy coping strategies, and is completed with the first three months post-injury.

DETAILED DESCRIPTION:
Although the majority of patients with mild traumatic brain injury (MTBI) experience complete recovery within three months, a sizeable group continues to report frequent and severe symptoms such as headaches, fatigue, difficulty concentrating, forgetfulness, and irritability, in what is labeled persistent post-concussion syndrome (PCS). Persistent PCS is associated with vocational, recreational, and social disability. Early education and reassurance (treatment as usual) is effective in general, but appears insufficient for this subgroup.

Recent research has identified risk factors for persistent PCS, including inaccurate illness beliefs, maladaptive coping behaviour, and emotional distress. The present study will evaluate the additive efficacy of a cognitive-behavioural therapy protocol designed to modify these risk factors, over and above treatment as usual.

Participants with MTBI will be recruited within six weeks of injury. Those identified as being at-risk for persistent PCS based on evidence-based criteria will receive treatment as usual and then be randomly assigned to receive either no further intervention or cognitive-behavioural therapy. We hypothesize that the group receiving cognitive-behavioural therapy will have fewer PCS symptoms and be less disabled at follow-up. We also hypothesize that compensation-seeking status will mitigate this improvement and that illness beliefs, coping behaviour, and emotional distress will mediate this improvement. A blinded rater will conduct the baseline and outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

* Incurred head trauma within six weeks of study entry
* Meet American Congress of Rehabilitation criteria for MTBI, documented by the referring/treating physician
* Subjective report at least one symptom attributable to head trauma
* English as preferred language for communication
* Considered at-risk for persistent PCS based on prognostic model from Whittaker et al. (2007)

Exclusion Criteria:

* Medical documentation of skull fracture or acute intracranial abnormality on neuroimaging, consistent with "mild-complicated" TBI
* Self-reported history of a neurological disorder (including prior MTBI within the past six months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
PCS symptoms (Rivermead Postconcussion Symptoms Questionnaire) | Pre-intervention and three months later
Functional disability (Mayo-Portland Participation Index) | Pre-intervention and three months later

SECONDARY OUTCOMES:
Illness beliefs (Illness Perceptions Questionnaire-Revised) | Pre-intervention and three months later
Coping style (PCS Coping Inventory) | Pre-intervention and three months later
Psychological distress (Hospital Anxiety and Depression Scale) ) | Pre-intervention and three months later
Pain (Brief Pain Scale) | Pre-intervention and three months later
Psychiatric diagnosis (MINI International Neuropsychiatric Interview) | Pre-intervention and three months later

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia; Brad Hallam, Study Director — University of British Columbia; Alice Rose, Study Director — Vancouver Coastal Health; Heather Underwood, Study Director — University of British Columbia; Allen Thornton, Study Director — Simon Fraser University; Kevin Whitfield, Study Director — Simon Fraser University; Maureen Whittal, Study Director — University of British Columbia
Locations (1):
- GF Strong Rehab Centre, 4255 Laurel Street, Vancouver, British Columbia, Canada